CLINICAL TRIAL: NCT00398905
Title: Controlled, Double-Blind, Randomised, Dose-Ranging Study on the Prevention of VTE in Patients Undergoing Elective Total Hip Replacement- ODIXa-HIP2 Study BAY 59-7939
Brief Title: Dose-Ranging Study of BAY 59-7939 on the Prevention of VTE in Patients Undergoing Elective Total Hip Replacement
Acronym: ODIXa-HIP2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Healthcare AG
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 10944
Record Dates: First submitted 2006-11-07; First posted 2006-11-14 (Estimated); Last update posted 2009-05-08 (Estimated); Status verified 2009-05

CONDITIONS: Venous Thromboembolism
Keywords: Prevention of venous thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (6):
- Arm 1 (Experimental)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Arm 2 (Experimental)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Arm 3 (Experimental)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Arm 4 (Experimental)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Arm 5 (Experimental)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Arm 6 (Active Comparator)
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — 2,5 mg twice daily (5 mg total daily dose)
  Arms: Arm 1
Drug: Rivaroxaban (Xarelto, BAY59-7939) — 5 mg twice daily (10 mg total daily dose)
  Arms: Arm 2
Drug: Rivaroxaban (Xarelto, BAY59-7939) — 10 mg twice daily (20 mg total daily dose)
  Arms: Arm 3
Drug: Rivaroxaban (Xarelto, BAY59-7939) — 20 mg twice daily (40 mg total daily dose)
  Arms: Arm 4
Drug: Rivaroxaban (Xarelto, BAY59-7939) — 30 mg twice daily (60 mg total daily dose)
  Arms: Arm 5
Drug: Enoxaparin — 40 mg once daily (40 mg total daily dose)
  Arms: Arm 6

SUMMARY:
Patients undergoing surgery, especially hip and knee surgery, are at high risk for VTE. The administration of drugs for thromboprophylaxis, such as heparins, significantly lowers that risk, but heparins have to be applied by injections below the skin. The purpose of this study was to compare the safety and efficacy of BAY 59-7939 with the safety and efficacy of the licensed drug enoxaparin and to find the optimal dose of BAY 59-7939 for the anticipated phase III trials. Enoxaparin, a so-called low molecular weight heparin, is approved and widely used in the area of thromboprophylaxis and was given once daily subcutaneously. In this study 5 different doses of the investigational drug BAY 59-7939 were tested in comparison to Enoxaparin. The following doses of BAY 59-7939 were tested: 2.5 mg twice daily (5 mg total daily dose); 5 mg twice daily (10 mg total daily dose), 10 mg twice daily (20 mg total daily dose), 20 mg twice daily (40 mg total daily dose) and 30 mg twice daily ( 60 mg total daily dose). This study ran for approximately 7 months in a number of countries. In total, 726 patients were enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18 years or above and postmenopausal female patients
* Patients scheduled for elective primary total hip replacement (cemented or non-cemented prosthesis
* Patients written informed consent for participation after receiving detailed written and oral previous information to any study specific procedures

Exclusion Criteria:

* Any VTE prior to randomization
* Myocardial infarction (MI) or TIA or ischaemic stroke within the last 6 months prior to randomisation
* History of heparin-induced thrombocytopenia, allergy to heparins
* Intracerebral or intraocular bleeding within the last 6 months prior to randomisation
* History of gastrointestinal disease with gastrointestinal bleeding within the last 6 months prior to the study
* History or presence of gastrointestinal disease which could result in an impaired absorption of the study drug (e.g. severe active inflammatory bowel disease, short gut syndrome)
* Amputation of one leg
* Heart insufficiency NYHA III-IV
* Congenital or acquired haemorrhagic diathesis (PT INR/aPTT not within normal limits) including patients with acquired or congenital thrombopathy
* Thrombocytopenia (platelets < 100.000/µl)
* Macroscopic haematuria.
* Allergy to contrast media.
* Severe hypertension (SBP > 200mmHg, DBP > 100 mmHg)
* Impaired liver function (transaminases > 2 x ULN)
* Impaired renal function (serum creatinine > 1.5 x ULN or creatinine clearance < 30 ml/min)
* Active malignant disease
* Presence of active peptic ulcer or gastrointestinal disease with increased risk of gastrointestinal bleeding
* Body weight < 45 kg
* Drug- or alcohol abuse
* Patients who cannot stop therapy ( in the opinion of the investigator/ physician) with anticoagulants (e.g. phenprocoumon, warfarin-sodium, heparins and factor Xa inhibitors other than study medication) and fibrinolytic therapy should be excluded from the study
* Therapy with acetylic salicylic acid or other thrombocyte aggregation inhibitors (e.g. clopidogrel, dipyridamole and ticlopidine) should be stopped one week before enrolment. Patients not able to stop ASA therapy will be excluded
* All other drugs influencing coagulation, (exception: NSAIDs with half life < 17 hrs will be allowed)
* Systemic and topical treatment with azole compounds (e.g. ketoconazole, fluconazole, itraconazole) and other strong CYP3A4 inhibitors e.g. HIV-protease inhibitors. Azole compounds and other strong CYP3A4 inhibitors
* Therapy with another investigational product within 30 days prior start of study
* Planned intermittent pneumatic compression during active treatment period
* Planned epidural anaesthesia with indwelling epidural catheter (spinal or epidural anaesthesia without indwelling catheter are allowed)
* Concomitant participation in another trial or study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 726 (Actual)
Dates: Start 2004-01; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Composite Endpoint: Any Deep Vein Thrombosis (DVT) (proximal and/or distal) and Non fatal Pulmonary Embolism (PE) and Death from all causes | 5-9 days after surgery

SECONDARY OUTCOMES:
Incidence of DVTs (total, proximal, distal) | 5-9 days after surgery
Incidence of symptomatic Venous Thrombo Embolisms (VTEs) | 5-9 days after surgery
Incidence of symptomatic VTEs (total, PE, DVT) within 30 days after stop of treatment with the study drug | 40 days
Healthcare Resource Utilisation Questionnaire | 9 days and 40 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (58):
- Austria (3):
  - Wiener Neustadt, Lower Austria
  - Linz, Upper Austria
  - Vienna, Vienna
- Belgium (5):
  - Baudour
  - Bruxelles - Brussel
  - Genk
  - Huy
  - Sint-Truiden
- Denmark (4):
  - Hellerup
  - Herlev
  - Hørsholm
  - Silkeborg
- France (3):
  - Amiens
  - Lille
  - Poitiers
- Germany (10):
  - Rheinfelden, Baden-Wurttemberg
  - Ulm, Baden-Wurttemberg
  - Fürth, Bavaria
  - Garmisch-Partenkirchen, Bavaria
  - Sommerfeld, Brandenburg
  - Frankfurt am Main, Hesse
  - Marburg, Hesse
  - Düsseldorf, North Rhine-Westphalia
  - Dresden, Saxony
  - Berlin, State of Berlin
- Israel (4):
  - Haifa
  - Tel Aviv
  - Tel Litwinsky
  - Ẕerifin
- Italy (7):
  - Rozzano, Milano
  - Gubbio, Perugia
  - Milan
  - Pavia
  - Perugia
  - Reggio Emilia
  - Varese
- Netherlands (3):
  - Hilversum
  - Nijmegen
  - Sittard
- Norway (5):
  - Bodø
  - Drammen
  - Notodden
  - Oslo
  - Rjukan
- Poland (6):
  - Bialystok
  - Gdansk
  - Krakow
  - Lodz
  - Lublin
  - Warsaw
- Spain (3):
  - Badalona, Barcelona
  - Barcelona, Barcelona
  - Valencia, Valencia
- Sweden (4):
  - Gothenburg
  - Halmstad
  - Jönköping
  - Kungälv
- London, Greater London, United Kingdom